CLINICAL TRIAL: NCT03494218
Title: Reliability and Validity of the Nociception Coma Scale (-Revised)-Chinese Version
Brief Title: Reliability and Validity of the NCS (NCS-R)-Chinese Version
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jing Wang, Dr, Hangzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2017R423055
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Minimally Conscious State; Vegetative State
Keywords: disorders of consciousness; vegetative state; minimally conscious state; consciousness; pain assessment; nociception test
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: The order of the administration was randomly selected. All patients' total scores assessed by rater A were recorded to test the internal consistency of NCS-R (A1). Meanwhile, to assess the concurrent validity, the scores of the FLACC were recorded together with NCS-R by rater A on day 1. In order to analyze the test-retest reliability, rater A complete the second evaluation of NCS-R on day 2 (A2)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vegetative state (Experimental): patients with vegetative state lack awareness of self and environment even in the presence for eye-opening and sleep-wake cycles using CRS-R. The nailbed pressure was applied for 5 seconds and ended as soon as the behavioral response were captured. The raters recorded patients' behavioral responses using Nociception Coma Scale (NCS) during 10 seconds after each noxious stimulus.
  Interventions: Diagnostic Test: Nociception Coma Scale (NCS)
- minimally conscious state (Experimental): Patients with minimally conscious state display inconsistent, but reproducible and discernible signs of awareness using CRS-R. The nailbed pressure was applied for 5 seconds and ended as soon as the behavioral response were captured. The raters recorded patients' behavioral responses using Nociception Coma Scale (NCS) during 10 seconds after each noxious stimulus.
  Interventions: Diagnostic Test: Nociception Coma Scale (NCS)

INTERVENTIONS:
Diagnostic Test: Nociception Coma Scale (NCS) — Patients have been assessed with both the Nociception Coma Scale (NCS) and the FLACC.
  Other Names: the Face Legs Activity Cry and Consolability (FLACC)

SUMMARY:
The aim of this study was to translate the NCS from English into Chinese and determine the validity of this Chinese version.

DETAILED DESCRIPTION:
The assessment and early diagnosis of pain is of great importance for pain management and treatment in patients with disorders of consciousness. The Nociception Coma Scale (- Revised) is only applicable to assess pain of DOC patients in international clinical setting. The aim of this study was to translate the NCS from English into Chinese and determine the validity of this Chinese version. To test internal reliability and inter-rater reliability, both rater A and rater B assess the perception of pain on day 1; and to obtain test-retest reliability, rater A assessed all patients repeatedly on day 2. 'Faces, Legs, Activity, Cry, Consolability' (FLACC) was used to analysis concurrent validity by rater A.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old;
* no administration of neuromuscular blockers or sedation within the 24 hours of enrolment;
* the presence of periods of eye opening (indicating wakefulness and rest cycles);
* a diagnosis of VS or MCS, based on more than 4 times behavioral assessment performed using the Coma Recovery Scale-Revised within 2 weeks.

Exclusion Criteria:

* Coma;
* documented history of prior brain injury;
* psychiatric or neurologic illness;
* neuromuscular blocking agents or sedative drugs administered within the prior 24 hours;
* no documented history of a prior coma, critical illness or unstable medical condition;
* upper limb contusions, fractures (based on the imaging examination) or flaccid paralysis (by using noxious stimuli to upper limbs, motor sub-scale scores <1).

Ages: 19 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
The level of perception of pain in DOC patients | Within 2 days
  This original NCS consists of four subscales to assess motor, verbal, visual and facial behavioral responses and each subscale score ranges from 0 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Di, Pro, Study Chair — International Vegetative State and Consciousness Science Institute, Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Chatelle C, Majerus S, Whyte J, Laureys S, Schnakers C. A sensitive scale to assess nociceptive pain in patients with disorders of consciousness. J Neurol Neurosurg Psychiatry. 2012 Dec;83(12):1233-7. doi: 10.1136/jnnp-2012-302987. Epub 2012 Aug 20. PMID 22906615